CLINICAL TRIAL: NCT04189055
Title: Cetuximab as Salvage Therapy in Patients With Neo Wild-type RAS/RAF Metastatic Colorectal Cancer With Liver Metastases. A Proof-of-concept Study
Brief Title: Cetuximab as Salvage Therapy in Patients With Neo Wild-type RAS/RAF Metastatic Colorectal Cancer With Liver Metastases.
Acronym: CETIDYL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Franco-Britannique-Fondation Cognacq-Jay (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FBH-001
Record Dates: First submitted 2019-11-27; First posted 2019-12-06 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Cancer Colorectal
Keywords: Liver metastasis; KRAS; NRAS
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort #1 (Experimental): Cetuximab monotherapy (500mg/m² IV, day 1)
  Interventions: Drug: Cetuximab
- Cohort #2 (Experimental): Cetuximab and irinotecan (cetuximab 500mg/m² IV, day 1; irinotecan 180mg/m² IV, day 1).
  Interventions: Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: Cetuximab — Cetuximab 500mg/m² IV, day 1
  Other Names: Erbitux
Drug: Irinotecan — Irinotecan 180mg/m² IV, day 1
  Other Names: Campto
  Arms: Cohort #2

SUMMARY:
The purpose of this study is to investigate the efficacy of cetuximab or cetuximab-irinotecan in patients with neo wild-type colorectal cancer who have been previously treated for metastatic disease.

Patients will be included in cohort #1 or cohort #2. The inclusion in cohort #2 will start when the results of the cohort #1 are available.

Patient will receive either cetuximab alone (cohort #1) or cetuximab with irinotecan (cohort #2).

DETAILED DESCRIPTION:
Background - Rationale

KRAS and NRAS mutations are present in roughly 50% of patients with advanced colorectal cancer and predict failure of anti-EGFR mabs therapies, thus genotyping colorectal cancer (CRC) is mandatory for personalized treatments.

Research has been selectively concentrated on the emergence of resistant clones in the blood of patients with wild-type (WT) RAS CRC as biomarker of anti-EGFR therapy resistance.

It has been suggested that patients with metastatic CRC harboring mutated primary tumors, thus not candidate to EGFR inhibitors, frequently have WT RAS circulating tumor cells in blood. Preliminary data suggest that patients with mutant KRAS colon cancer can frequently (50%) switch to a prevalent WT KRAS disease in course of treatment with anti-angiogenic drugs.

In patients with RAS wild-type colorectal cancer who previously received standard therapies, anti-EGFR mabs achieve a response rate of 20% as monotherapy and 30-40% in combination with irinotecan.

The aim of this study is to evaluate the efficacy of cetuximab in patients with pretreated neo wild-type colorectal cancer using liquid biopsies for RAS molecular assessment

Study Objectives

Primary:

• To evaluate the response rate using RECIST 1.1

Secondary:

* To evaluate progression-free survival (PFS), overall survival (OS)
* To evaluate disease control rate (DCR)
* To evaluate safety

Exploratory:

* Frequency of neo wild-type tumors
* Frequency of RAS and BRAF neomutations during treatment

Study Design Prospective multicentric single-arm open-label phase II study in to 2 successive patient cohorts (cohort #1 followed by cohort #2).

Molecular screening using Idylla™ (Biocartis) ctKRAS and ctNRAS/BRAF Mutation Assays.

Cohort #1: Patients will be treated with cetuximab monotherapy (cetuximab 500mg/m² IV, day 1).

Cohort #2: Patients will be treated with cetuximab and irinotecan (cetuximab 500mg/m² IV, day 1; irinotecan 180mg/m² IV, day 1).

In both cohorts, treatment will be given intravenously every 14 days (q2w) until disease progression or limiting toxicity. Tumor evaluations will be done with CT-scan (or MRI) every 8 weeks using RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent and stated willingness to comply with all study procedures and availability for the duration of the study,
2. Male or female subjects, ≥18 years of age,
3. ECOG performance status (ECOG PS, Appendix 15.1) ≤2,
4. Unresectable metastatic RAS mutant (either KRAS or NRAS tumor gene mutation) colorectal cancer,
5. At least one (≥1) measurable and/or evaluable liver metastasis,
6. Prior therapy (resistant or intolerant) with fluoropyrimidines, oxaliplatin, irinotecan and antiangiogenic agent (ie, bevacizumab and/or aflibercept),
7. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

   Hematological status: neutrophils (ANC) ≥1.5x109/L; platelets ≥100x109/L; haemoglobin ≥9g/dL Adequate renal function: serum creatinine clearance (MDRD) ≥ 50 mL/min/1,73 m2 Adequate liver function: serum bilirubin ≤1.5x upper normal limit (ULN), alkaline phosphatase <5xULN, AST and ALT ≤5xULN, Adequate serum electrolyte levels (magnesium, potassium, calcium) prior to initiation of study treatment,
8. Negative pregnancy test within 7 days prior to initiation of the study drug for female patients of childbearing potential,
9. Effective contraception for both male and female subjects if the risk of conception exists
10. Registration in a national health care system.

Exclusion Criteria:

1. Known allergy or hypersensitivity reactions to any study drug,
2. Women who are pregnant or breastfeeding,
3. Inability to comply with study and follow-up procedures as judged by the Investigator,
4. Patient with BRAF mutant colorectal cancer
5. History of interstitial lung disease
6. Treatment with strong CYP3A4-enzyme inducers such as anticonvulsants (phenytoin, phenobarbital or carbamazepine), rifampin, rifabutin and St. John's wort for patients of cohort #2
7. Treatment with strong CYP3A4-enzyme inhibitors (e.g. grapefruit juice, clarithromycin, indinavir, itraconazole, lopinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telaprevir, voriconazole) for patients of cohort #2
8. Treatment with strong UGT1A inhibitors (e.g. atazanavir, gemfibrozil, indinavir) for patients of cohort # 2
9. Patients of cohort #2 with known UGT1A deficiency
10. Uncontrolled illness, including but not limited to ongoing bacterial, viral or fungal infection requiring systemic therapy, metabolic dysfunction, physical examination/ clinical laboratory finding that leads to a reasonable suspicion of a disease/condition that contraindicates the use of any of investigational drugs that may affect the interpretation of the results, or that may render the subject at high risk of treatment complications.
11. Patient with current intestinal obstruction or history of chronic inflammatory bowel disease
12. Subjects under guardianship, curatorship or judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
response rate | 4 months
  Tumor measurements will be obtained at baseline and every 8 weeks following treatment initiation. At the investigator's discretion, tumor assessments may be repeated at any time if progressive disease is suspected. Tumor response and progression will be assessed by the Investigator using RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival | time interval from inclusion to the date of death from any cause. Assessed up to 12 months after the beginning of the study
  OS is defined as the time interval from the date of inclusion to the date of death from any cause. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period.
Progression-free survival | the time interval from inclusion to the date of first documented disease progression or death from any cause, whichever occurs first. Assessed up to 12 months after the beginning of the study
  PFS is defined as the time interval from the date of inclusion to the date of first documented disease progression or death from any cause, whichever occurs first. Alive patients without progression will be censored at the last tumor assessment, either during study treatment period or during follow-up period.
Disease Control rate | from baseline until end of treatment, assessed up to 12 months after the beginning of the study
  Disease control rate (DCR) is defined as the percentage of patients achieving CR, PR, or stable disease (SD).
Tolerance | Assessed from study entry to 1 month after last study drug administration, assessed up to 12 months after the beginning of the study
  Frequency of adverse events using NCI-CTCAE v5.0

OTHER OUTCOMES:
Tumor biomarkers | Assessed from study entry to end of study treatment, assessed up to 12 months after the beginning of the study
  Tumor biomarkers will be tested : mismatch repair system (pMMR vs dMMR), HER1 (EGFR expression), HER2 expression, amphiregulin (AREG) and HER1 (EGFR GCN, cut-off 4.0), HER2, PI3KCA, PTEN, IRS2,

CONTACTS AND LOCATIONS:
Overall Officials: Benoist CHIBAUDEL, MD, Principal Investigator — Franco-British Hospital - GCS IHFB Cognacq-Jay
Locations (1):
- Franco-British Hospital - GCS IHFB Cognacq-Jay, Levallois-Perret, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amado RG, Wolf M, Peeters M, Van Cutsem E, Siena S, Freeman DJ, Juan T, Sikorski R, Suggs S, Radinsky R, Patterson SD, Chang DD. Wild-type KRAS is required for panitumumab efficacy in patients with metastatic colorectal cancer. J Clin Oncol. 2008 Apr 1;26(10):1626-34. doi: 10.1200/JCO.2007.14.7116. Epub 2008 Mar 3. PMID 18316791
- [Background] Andre T, Blons H, Mabro M, Chibaudel B, Bachet JB, Tournigand C, Bennamoun M, Artru P, Nguyen S, Ebenezer C, Aissat N, Cayre A, Penault-Llorca F, Laurent-Puig P, de Gramont A; GERCOR. Panitumumab combined with irinotecan for patients with KRAS wild-type metastatic colorectal cancer refractory to standard chemotherapy: a GERCOR efficacy, tolerance, and translational molecular study. Ann Oncol. 2013 Feb;24(2):412-419. doi: 10.1093/annonc/mds465. Epub 2012 Oct 5. PMID 23041588
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Background] Elez E, Kocakova I, Hohler T, Martens UM, Bokemeyer C, Van Cutsem E, Melichar B, Smakal M, Csoszi T, Topuzov E, Orlova R, Tjulandin S, Rivera F, Straub J, Bruns R, Quaratino S, Tabernero J. Abituzumab combined with cetuximab plus irinotecan versus cetuximab plus irinotecan alone for patients with KRAS wild-type metastatic colorectal cancer: the randomised phase I/II POSEIDON trial. Ann Oncol. 2015 Jan;26(1):132-140. doi: 10.1093/annonc/mdu474. Epub 2014 Oct 15. PMID 25319061
- [Background] Hecht JR, Patnaik A, Berlin J, Venook A, Malik I, Tchekmedyian S, Navale L, Amado RG, Meropol NJ. Panitumumab monotherapy in patients with previously treated metastatic colorectal cancer. Cancer. 2007 Sep 1;110(5):980-8. doi: 10.1002/cncr.22915. PMID 17671985
- [Background] Jonker DJ, O'Callaghan CJ, Karapetis CS, Zalcberg JR, Tu D, Au HJ, Berry SR, Krahn M, Price T, Simes RJ, Tebbutt NC, van Hazel G, Wierzbicki R, Langer C, Moore MJ. Cetuximab for the treatment of colorectal cancer. N Engl J Med. 2007 Nov 15;357(20):2040-8. doi: 10.1056/NEJMoa071834. PMID 18003960
- [Background] Karapetis CS, Khambata-Ford S, Jonker DJ, O'Callaghan CJ, Tu D, Tebbutt NC, Simes RJ, Chalchal H, Shapiro JD, Robitaille S, Price TJ, Shepherd L, Au HJ, Langer C, Moore MJ, Zalcberg JR. K-ras mutations and benefit from cetuximab in advanced colorectal cancer. N Engl J Med. 2008 Oct 23;359(17):1757-65. doi: 10.1056/NEJMoa0804385. PMID 18946061
- [Background] Pfeiffer P, Nielsen D, Bjerregaard J, Qvortrup C, Yilmaz M, Jensen B. Biweekly cetuximab and irinotecan as third-line therapy in patients with advanced colorectal cancer after failure to irinotecan, oxaliplatin and 5-fluorouracil. Ann Oncol. 2008 Jun;19(6):1141-5. doi: 10.1093/annonc/mdn020. Epub 2008 Feb 14. PMID 18281264